CLINICAL TRIAL: NCT04625634
Title: Simulation of Consecutive Day Shift Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Riana Pryor, Primary Investigator, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00003948
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Hyperthermia; Fatigue; Heat
MeSH Terms: conditions — Hyperthermia; Heat Stress Disorders

STUDY DESIGN:
Intervention Model Description: Repeated measures study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Consecutive work (Experimental): Subjects will complete 2 consecutive days of simulated firefighting tasks in the heat. The simulated work consists of 20 minutes of simulated structural work in a hot environment, followed by 20 minutes of seated rest in a temperate room, mimicking a typical recovery period in structural firefighting. Subjects then re-enter the environmental chamber and complete 23 minutes of simulated overhaul work in a temperate environment.
  Interventions: Other: 2 days of work heat stress

INTERVENTIONS:
Other: 2 days of work heat stress — 2 consecutive days of identical simulated structural firefighting tasks.

SUMMARY:
The purpose of this study is to determine differences in physiological recovery between two consecutive days of simulated fire suppression work. The secondary purpose is to determine differences in heat gain and heat loss between two consecutive days of simulated fire suppression work. Subjects will complete two consecutive days of simulated structural firefighting shift work, 24 hours apart. Before and after each laboratory visit, subjects will continuously wear a Holter monitor and ambulatory blood pressure monitor to quantify parasympathetic tone and recovery from work.

ELIGIBILITY:
Inclusion Criteria:

* 18-39 y old men and women
* Self-reported to be healthy

Exclusion Criteria:

* History of any cardiovascular, neurologic, renal, or metabolic disease
* Current tobacco use or regular use within the last 2 years
* Taking medications with known thermoregulatory or cardiovascular effects (e.g., aspirin, acetaminophen, ibuprofen, beta blockers, diuretics, psychotropics, etc.)
* History of exertional heat stroke
* Currently pregnant or breastfeeding, or planning to become pregnant during the study
* Inability to follow the rules of the protocols or understand the consent form
* No contraindications for ingestion of the gastrointestinal temperature pill

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Core temperature | 20 minutes
  Gastrointestinal temperature measured with an ingestable pill.
Heart rate | 20 minutes
  Heart rate measured with a wearable heart rate strap and monitor

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Research and Exercise in Special Environments, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual data can be made available upon written request.